CLINICAL TRIAL: NCT04019873
Title: 'COMBINE-2': Real-world Evidence for Effectiveness of Two Drug Regimen, Antiretroviral Therapy With Integrase Inhibitors Plus a Reverse Transcriptase Inhibitor
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 207859
Record Dates: First submitted 2018-07-19; First posted 2019-07-15 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: 2DR; HIV; Lamivudine; COMBINE-2; Dolutegravir
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment-naïve participants: Participants received a two-drug regimen (2DR) consisting of an integrase inhibitor plus a reverse transcriptase inhibitor, as a first-line treatment for Human Immunodeficiency Virus (HIV) infection.
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC); Drug: Rilpivirine (RPV)
- Stable switch participants: Participants received a two-drug regimen (2DR) consisting of an integrase inhibitor plus a reverse transcriptase inhibitor, as a switching treatment option for HIV infection, whilst virologically suppressed (whilst having HIV RNA suppression) on current treatment.
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC); Drug: Rilpivirine (RPV)
- Prior virological failure participants: Participants received a two-drug regimen (2DR) consisting of an integrase inhibitor plus a reverse transcriptase inhibitor, as a second-line treatment for HIV infection, due to virological failure (VF) on prior treatment.
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC); Drug: Rilpivirine (RPV)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — DTG is a 2nd generation integrase strand transfer inhibitor. Subjects receiving DTG as a part of 2DR treatment will be included in the study.
Drug: Lamivudine (3TC) — 3TC is a nucleoside reverse transcriptase inhibitor. Subjects receiving 3TC as a part of 2DR treatment will be included in the study.
Drug: Rilpivirine (RPV) — RPV is a non-nucleoside reverse transcriptase inhibitor. Subjects receiving RPV as part of 2DR treatment will be included in the study.

SUMMARY:
Dolutegravir (DTG) is a well-tolerated 2nd generation integrase strand transfer inhibitor (INSTI); rilpivirine (RPV) is a well-tolerated non- nucleoside reverse transcriptase inhibitors (NNRTI) and lamivudine (3TC) is a nucleoside reverse transcriptase inhibitors (NRTIs). This study aims to gather the real-world evidence to evaluate effectiveness of the two-drug regimen (2DR). This is a multi-site observational study in subjects who have started and/or who plan to initiate 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor. The study does not require any changes to the routine standard of care that subjects receive. Approximately 500 eligible subjects will be included from potential investigational sites across Europe and data from them will be collected either retrospectively or prospectively.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive male or female subjects aged 18 years or over and who have started 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor from 2014 onwards as a first-line treatment among naïve subjects, or a switching option for those with HIV RNA suppression on current treatment (stable switches), or a second-line treatment for those with virological failure on prior treatment.

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of HIV positive male or female subjects aged 18 years or over and who have started 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor from 2014 onwards as a first-line treatment among naïve subjects, or a switching option for those with HIV RNA suppression on current treatment (stable switches), or a second-line treatment for those with virological failure on prior treatment.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Started | 23 | 735 | 16
Completed | 22 | 696 | 14
Not Completed | 1 | 39 | 2
Not completed — Discontinued from the treatment | 1 | 39 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment-naïve Participants: Participants received a two-drug regimen (2DR) consisting of an integrase inhibitor plus a reverse transcriptase inhibitor, as a first-line treatment for HIV infection.
- Total: Total of all reporting groups
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants | Total
Number analyzed (Participants) | 23 | 735 | 16 | 774
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 37 [34 to 53] | 54 [47 to 59] | 57 [51 to 61] | 53 [47 to 59]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 19 | 556 | 13 | 588
  Female | 3 | 176 | 3 | 182
  Transgender | 1 | 2 | 0 | 3
  Other, Unspecified | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 492 | 12 | 520
  Black | 1 | 140 | 3 | 144
  Asian | 0 | 8 | 1 | 9
  Other, unspecified | 6 | 95 | 0 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-naïve Participants With Human Immunodeficiency Virus Ribonucleic Acid (HIV-RNA) Levels Less Than (<)50 Copies/Milliliter (c/mL) at 24 Weeks After 2DR (Two-drug Regimen) Initiation
Time Frame: At Week 24
Population: Analysis population included only the Treatment-naïve participants who had a viral load (VL) measurement at the specified time point (at the 24-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 20
Participants | 19

2. Primary Outcome: Number of Treatment-naïve Participants With HIV-RNA Levels <50 c/mL at 48 Weeks After 2DR Initiation
Time Frame: At Week 48
Population: Analysis population included only the Treatment-naïve participants who had a viral load (VL) measurement at the specified time point (at the 48-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 19
Participants | 19

3. Primary Outcome: Number of Treatment-naïve Participants With HIV-RNA Levels <50 c/mL at 96 Weeks After 2DR Initiation
Time Frame: At Week 96
Population: Analysis population included only the Treatment-naïve participants who had a viral load (VL) measurement at the specified time point (at the 96-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 20
Participants | 20

4. Primary Outcome: Number of Treatment-experienced Viremic Participants With HIV-RNA Levels <50 c/mL at Week 24
Time Frame: At Week 24
Population: Analysis population included only the Prior virological failure participants who had a viral load (VL) measurement at the specified time point (at the 24-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 16
Participants | 14

5. Primary Outcome: Number of Treatment-experienced Viremic Participants With HIV-RNA Levels <50 c/mL at Week 48
Time Frame: At Week 48
Population: Analysis population included only the Prior virological failure participants who had a viral load (VL) measurement at the specified time point (at the 48-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 12
Participants | 11

6. Primary Outcome: Number of Treatment-experienced Viremic Participants With HIV-RNA Levels <50 c/mL at Week 96
Time Frame: At Week 96
Population: Analysis population included only the Prior virological failure participants who had a viral load (VL) measurement at the specified time point (at the 96-week time point). Stable switch participants were not included in the analysis, as these participants were already suppressed (HIV RNA <50 c/mL) at baseline. Per the protocol, the primary endpoints of suppression at 24, 48, and 96 weeks were only evaluated for Treatment-naïve participants and Prior virological failure participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 12
Participants | 10

7. Primary Outcome: Number of Treatment-naïve Participants Experiencing Virologic Failure (VF) [Up to 24 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA level greater than or equal to [>=] 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL>=200 copies/mL after at least 24 weeks of treatment).
Time Frame: Up to 24 weeks
Population: Analysis population included all the individuals, (among the Treatment-naïve participants) who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment for HIV infection, and who had at least one VL measurement up to the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 23
Participants | 0

8. Primary Outcome: Number of Treatment-naïve Participants Experiencing VF [Up to 48 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA level greater than or equal to [>=] 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL>=200 copies/mL after at least 48 weeks of treatment).
Time Frame: Up to 48 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 23
Participants | 0

9. Primary Outcome: Number of Treatment-naïve Participants Experiencing VF [Up to 96 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA level greater than or equal to [>=] 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL>=200 copies/mL after at least 96 weeks of treatment).
Time Frame: Up to 96 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants
Number analyzed (Participants) | 23
Participants | 0

10. Primary Outcome: Number of Stable Switch Participants With VF Within the First 24 Weeks
Description: VF was defined as 2 consecutive HIV RNA >=50 c/mL or 1 HIV RNA >50c/mL followed by study treatment discontinuation or missing value.
Time Frame: Up to Week 24
Population: Analysis population included all the individuals, (among the Stable switch participants) who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period (as a switching treatment option for HIV infection, whilst virologically suppressed on current treatment) and who had a VL measurement up to the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Switch Participants
Number analyzed (Participants) | 735
Participants | 1

11. Primary Outcome: Number of Stable Switch Participants With VF Within the First 48 Weeks
Description: as for outcome 10
Time Frame: Up to Week 48
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Switch Participants
Number analyzed (Participants) | 735
Participants | 3

12. Primary Outcome: Number of Stable Switch Participants With VF Within the First 96 Weeks
Description: as for outcome 10
Time Frame: Up to Week 96
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Switch Participants
Number analyzed (Participants) | 735
Participants | 10

13. Primary Outcome: Number of Treatment-experienced Viremic Participants Experiencing VF [Up to 24 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA >= 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL >=200 copies/mL after at least 24 weeks of treatment). Treatment-experienced viremic participants refers to individuals who have previously undergone HIV treatment but had virological failure in prior treatment.
Time Frame: Up to 24 weeks
Population: Analysis population included all the individuals, among the Prior virological failure participants, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a second-line treatment, due to VF on prior treatment, and who had a VL measurement up to the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 16
Participants | 0

14. Primary Outcome: Number of Treatment-experienced Viremic Participants Experiencing VF [Up to 48 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA >= 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL >=200 copies/mL after at least 48 weeks of treatment). Treatment-experienced viremic participants refers to individuals who have previously undergone HIV treatment but had virological failure in prior treatment.
Time Frame: Up to 48 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 16
Participants | 1

15. Primary Outcome: Number of Treatment-experienced Viremic Participants Experiencing VF [Up to 96 Weeks]
Description: VF was defined as virologic rebound (after achieving suppression, 2 consecutive HIV RNA >= 50 copies/mL or 1 HIV RNA level >=50 copies/mL followed by study treatment discontinuation) or virologic non-response (2 consecutive VL >=200 copies/mL after at least 96 weeks of treatment). Treatment-experienced viremic participants refers to individuals who have previously undergone HIV treatment but had virological failure in prior treatment.
Time Frame: Up to 96 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Virological Failure Participants
Number analyzed (Participants) | 16
Participants | 3

16. Secondary Outcome: Number of Participants With HIV RNA Levels >=200 c/mL After 24 Weeks, 48 Weeks and 96 Weeks
Time Frame: At Week 24, Week 48 and Week 96
Population: Analysis population included (only) the individuals, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment, or as a switching treatment option whilst virologically suppressed on current treatment, or as a second-line treatment, due to VF on prior treatment, and who had a VL measurement at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 20 | 735 | 16
Participants
  At 24 weeks | 0 | 1 | 2
  At 48 weeks: number analyzed (Participants) | 19 | 712 | 12
  At 48 weeks | 0 | 1 | 1
  At 96 weeks: number analyzed (Participants) | 20 | 574 | 12
  At 96 weeks | 0 | 2 | 1

17. Secondary Outcome: Number of Participants With Low Level Viremia
Description: Low level viremia was defined as virologic load >=50 and <200 c/mL.
Time Frame: At Week 24, Week 48 and Week 96
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 20 | 735 | 16
Participants
  At 24 weeks | 1 | 6 | 0
  At 48 weeks: number analyzed (Participants) | 19 | 712 | 12
  At 48 weeks | 0 | 8 | 0
  At 96 weeks: number analyzed (Participants) | 20 | 574 | 12
  At 96 weeks | 0 | 5 | 1

18. Secondary Outcome: Time to Virologic Suppression Among Treatment-naïve Participants and Treatment-experienced Viremic Participants, Who Achieved Suppression
Description: Suppression of VL was evaluated at 24 weeks, 48 weeks and 96 weeks and time to virologic suppression was planned to be evaluated until 96 weeks.
Time Frame: Up to Week 96
Population: Number of participants analyzed (N=23, 15) signifies participants who were evaluable for this outcome measure. As pre-specified in the protocol, a total of at least 90 treatment-naïve participants and 90 prior virologic failure participants should have been included for the power calculation of this endpoint.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Treatment-naïve Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 15
Months | NA [NA to NA] — NA signifies that median, lower and upper limit could not be estimated due to insufficient number of participants with events for fulfilling the power calculations. Data was used only for the descriptive purposes. | NA [NA to NA] — NA signifies that median, lower and upper limit could not be estimated due to insufficient number of participants with events for fulfilling the power calculations. Data was used only for the descriptive purposes.

19. Secondary Outcome: Time to Virologic Failure in the Stable Switch Population
Description: as for outcome 8
Time Frame: Up to Week 96
Population: Number of participants analyzed (N=10) signifies participants who were evaluable for this outcome measure. As pre-specified in the protocol, a total of at least 320 stable switch participants should have been included for the power calculation of this endpoint.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Stable Switch Participants
Number analyzed (Participants) | 10
Months | NA [NA to NA] — NA signifies that median, lower and upper limit could not be estimated due to insufficient number of participants with events for fulfilling the power calculations. Data was used only for the descriptive purposes.

20. Secondary Outcome: Number of Participants With Emergent Resistance Mutations Following Virologic Failure (VF) Events
Time Frame: Up to Week 96
Population: Analysis population included (only) the individuals,who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment,or as a switching treatment option whilst virologically suppressed on current treatment, or as a second-line treatment, due to VF on prior treatment, and who had a VL measurement at the specified time points. No participants had emergent resistance mutations following VF events
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 735 | 16
Participants | 0 | 0 | 0

21. Secondary Outcome: Number of Participants Who Discontinue Their Baseline 2DR and Who Stable Switch to a Different Regimen While Virologically Suppressed (HIV RNA <50 Copies/mL) at Switch
Description: A stable switch was defined as a switching option for participants with HIV RNA suppression on current treatment with viral load <50 c/mL at time of switch.
Time Frame: Up to Week 96
Population: Analysis population included all the individuals, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment, or as a switching treatment option whilst virologically suppressed on current treatment, or as a second-line treatment, due to VF on prior treatment, and who had at least one VL measurement up to the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 735 | 16
Participants | 1 | 35 | 1

22. Secondary Outcome: Number of Participants Who Discontinue Their Baseline 2DR and Who Switch Following Virologic Failure
Description: Virologic rebound or virologic non-response in participants, was considered as virologic failure.
Time Frame: Up to Week 96
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 735 | 16
Participants | 0 | 4 | 1

23. Secondary Outcome: Number of Participants Who Discontinue Their Baseline 2DR Who Are Switching for Safety or Other Reasons
Description: Safety reasons include tolerability, toxicity and other reasons.
Time Frame: Up to Week 96
Population: Analysis population included all the individuals, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment, or as a switching treatment option whilst virologically suppressed on current treatment, or as a second-line treatment, due to VF on prior treatment and had safety data collected in terms of drug related adverse events (AEs) and serious adverse events (SAEs) since first starting 2DR treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 735 | 16
Participants | 1 | 33 | 1

24. Secondary Outcome: Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward event resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Determination of an event as AE or SAE was at the discretion of the treating clinician and taken from the medical record.
Time Frame: Up to Week 96
Population: Analysis population included all the individuals, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period and had safety data collected in terms of drug related AEs and SAEs since first starting 2DR treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 23 | 735 | 16
Participants
  AEs | 1 | 39 | 1
  SAEs | 1 | 2 | 0

25. Secondary Outcome: Cluster of Differentiation (CD)4+ and CD8+ T Cell Counts
Time Frame: At baseline (Week 0), Week 24, Week 48 and Week 96
Population: Analysis population included only the individuals, who had initiated a 2DR with an integrase inhibitor plus a reverse transcriptase inhibitor prior to or during the study period, as a first-line treatment, or as a switching treatment option whilst virologically suppressed on current treatment, or as a second-line treatment, due to VF on prior treatment and who had immunological data collected since first starting 2DR treatment.
Measure: Median (Inter-Quartile Range); unit: cells per cubic millimeter (cells/mm^3)
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 17 | 509 | 13
cells per cubic millimeter (cells/mm^3)
  CD4 Count, Week 0 | 411 [340 to 553] | 684 [534 to 920] | 674 [523 to 807]
  CD4 Count, Week 24: number analyzed (Participants) | 15 | 353 | 12
  CD4 Count, Week 24 | 579 [477 to 693] | 712 [534 to 956] | 709 [541 to 980]
  CD4 Count, Week 48: number analyzed (Participants) | 11 | 358 | 11
  CD4 Count, Week 48 | 634 [465 to 976] | 709 [520 to 921] | 801 [576 to 883]
  CD4 Count, Week 96: number analyzed (Participants) | 13 | 460 | 11
  CD4 Count, Week 96 | 741 [610 to 1033] | 694 [528 to 898] | 804 [505 to 1151]
  CD8 Count, Week 0: number analyzed (Participants) | 10 | 486 | 13
  CD8 Count, Week 0 | 875 [677 to 1914] | 798 [585 to 1046] | 1015 [744 to 1179]
  CD8 Count, Week 24: number analyzed (Participants) | 9 | 343 | 12
  CD8 Count, Week 24 | 709 [564 to 812] | 796 [587 to 1118] | 879 [645 to 1396]
  CD8 Count, Week 48: number analyzed (Participants) | 6 | 347 | 11
  CD8 Count, Week 48 | 688 [661 to 1804] | 794 [586 to 1027] | 879 [640 to 1171]
  CD8 Count, Week 96: number analyzed (Participants) | 6 | 450 | 11
  CD8 Count, Week 96 | 1548 [930 to 2162] | 786 [558 to 1033] | 932 [760 to 1260]

26. Secondary Outcome: CD4/CD8 Ratio
Time Frame: At baseline (Week 0), Week 24, Week 48 and Week 96
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
Number analyzed (Participants) | 10 | 486 | 13
Ratio
  CD4/CD8, Week 0 | 0.60 [0.41 to 0.88] | 0.88 [0.61 to 1.24] | 0.72 [0.36 to 0.90]
  CD4/CD8, Week 24: number analyzed (Participants) | 9 | 343 | 12
  CD4/CD8, Week 24 | 0.72 [0.66 to 1.06] | 0.89 [0.66 to 1.28] | 0.75 [0.43 to 1.31]
  CD4/CD8, Week 48: number analyzed (Participants) | 6 | 347 | 11
  CD4/CD8, Week 48 | 1.02 [0.70 to 1.38] | 0.89 [0.64 to 1.24] | 0.90 [0.39 to 1.50]
  CD4/CD8, Week 96: number analyzed (Participants) | 6 | 450 | 11
  CD4/CD8, Week 96 | 0.79 [0.54 to 1.06] | 0.95 [0.65 to 1.29] | 0.95 [0.52 to 1.52]

ADVERSE EVENTS:
Time Frame: Non-serious AEs and serious AEs were collected from the day of the first exposure to the 2DR (date when 2DR was prescribed) until week 96, or at the earliest of the following events: date of last study contact, date of 2DR treatment discontinuation (except if the participant was switched to another 2DR), or the date of lost to follow-up.
Description: Serious and non-serious AEs reported in this module are presented under general disorders organ system classification as they were not classified initially by the physician during adverse events collection through the study.
Arm/Group | Treatment-naïve Participants | Stable Switch Participants | Prior Virological Failure Participants
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/735 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/735 | 0/16
Other Adverse Events (participants affected / at risk) | 1/23 | 39/735 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-naïve Participants (N=23) | Stable Switch Participants (N=735) | Prior Virological Failure Participants (N=16)
Low mood (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety and depression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nodding head syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-naïve Participants (N=23) | Stable Switch Participants (N=735) | Prior Virological Failure Participants (N=16)
Weight gain (General disorders) | 0 (0) | 8 (8) | 0 (0)
Diarrhea (General disorders) | 0 (0) | 3 (3) | 0 (0)
Sleep disorders (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (General disorders) | 0 (0) | 2 (2) | 0 (0)
Acute urinary retention (General disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety and depression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral flank pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
CNS AE (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cramps (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cytolisis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Destructive behaviour (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema of the lower limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulency (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercreatininaemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney function decline EGFR 58ML/MIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
Left leg numbness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Liquid stool (General disorders) | 0 (0) | 1 (1) | 0 (0)
Loose stools (General disorders) | 0 (0) | 1 (1) | 0 (0)
Low mood (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturnal and diurnal cough (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pantoprazolo (General disorders) | 0 (0) | 1 (1) | 0 (0)
Psychological problems and insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Right hand paresthesia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sweating (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tinitus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of gastroesophageal reflux (General disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of Parkinson disease (General disorders) | 0 (0) | 1 (1) | 0 (0)
Restless sleep (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vivid dreams (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04019873/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT04019873/SAP_001.pdf